CLINICAL TRIAL: NCT06164106
Title: Feasibility Trial of a Single Session of Crisis Response Planning for Youth at High Risk for Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Stephanie M Gorka, PhD, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023B0257
Record Dates: First submitted 2023-11-09; First posted 2023-12-11 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Suicide Prevention
Keywords: Suicide; Crisis Response Planning; Ecological Momentary Assessments
MeSH Terms: conditions — Suicide Prevention; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Crisis Response Planning (Experimental): The virtual crisis response planning (CRP) session will last between 30 minutes to 1-hour and be conducted via doxy.me with a trained study therapist. The virtual CRP is primarily text-based, instead of verbal, and utilizes the chat feature on doxy.me. CRP involves the following standard suicide intervention strategies: supportive listening, provision of crisis resources, and referral to a mental health professional (if not already established). The CRP active component involves a collaborative process in which the therapist invites the participant to share the events, symptoms, and contextual factors leading up to and surrounding their suicidal crisis. Next, the participant identifies their personal warning signs, self-management coping skills, reasons for living, and sources of social support. The participant types the components on a template via the white board feature on doxy.me. The CRP will be saved and serve as a concrete reference for participants in the real-world.
  Interventions: Behavioral: Virtual Crisis Response Planning
- In-Person Crisis Response Planning (Active Comparator): The in-person crisis response planning (CRP) session will last between 30 minutes to 1-hour. The in-person CRP will follow the same protocol and include the same treatment components as the virtual CRP. However, it will occur face-to-face, instead of on doxy.me, with a trained study therapist. The treatment components, outlined under the virtual CRP arm description, are written by the participant on an index card. The index card serves as a concrete reference for participants in the real-world.
  Interventions: Behavioral: In-Person Crisis Response Planning
- Virtual Crisis Risk Counseling (Active Comparator): The crisis risk counseling session will last between 30 minutes to 1-hour. It will occur virtually on doxy.me with a trained study therapist. It will include the following standard suicide intervention strategies: supportive listening, provision of crisis resources, and referral to a mental health professional (if not already established). The therapist will conduct a semi-structured suicide risk assessment interview, after which participants will complete a self-guided safety plan worksheet via the white board feature. The worksheet will take approximately 10-minutes to complete and will be done independently.
  Interventions: Behavioral: Crisis Risk Counseling

INTERVENTIONS:
Behavioral: Virtual Crisis Response Planning — Individuals complete a chat-based experimental collaborative suicide intervention virtually.
  Arms: Virtual Crisis Response Planning
Behavioral: In-Person Crisis Response Planning — Individuals complete a collaborative suicide intervention in-person.
  Arms: In-Person Crisis Response Planning
Behavioral: Crisis Risk Counseling — Individuals complete a standard crisis risk management intervention.
  Arms: Virtual Crisis Risk Counseling

SUMMARY:
The current study is a clinical trial, meaning a research study in which human subjects are prospectively assigned to one or more interventions to evaluate the effects of those interventions on health-related behavioral outcomes. Specifically, male and female adolescents with current suicidal intent will be randomly assigned to receive either a 1-hour session of virtual crisis response planning (CRP), a 1-hour session of in-person CRP, or a 1-hour session of standard crisis risk management (treatment as usual). The feasibility and acceptability of the virtual CRP, compared to in-person CRP, will be assessed 14 days post-treatment. Additional assessments of changes in mood, behavior, and suicidality will be collected daily for 14 days post-treatment via ecological momentary assessments. The investigators hypothesize the following: 1) Virtual CRP will be rated as more feasible and acceptable compared to traditional CRP and treatment as usual interventions; 2) Both versions of CRP will be associated with changes in frequency and severity of suicidal ideation and behavior compared to treatment as usual; 3) Virtual CRP will be equally as effective as traditional CRP at reducing suicide risk, suggesting that virtual CRP is a promising scalable intervention adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 14-18 years old at the time of assent/consent
* Participant's legal guardian is willing and able to give parental permission (if 14-17 years old)
* Participant is able to give informed assent or consent (as applicable by age)
* Participant endorses current desires to make a suicide attempt as defined as answering "yes" to item #3 on the Ask Suicide Screening Question (ASQ) tool

Exclusion Criteria:

* Factors that would interfere with data interpretation including serious medical or neurologic conditions
* Presence of current moderate to severe substance use disorder
* Lack of access to a personal smartphone
* Lack of fluency in English

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the experimental treatment as measured by ecological momentary assessments. | EMA surveys will be sent 5 times daily for 14 days post-intervention.
  Self-reported utilization of the crisis response planning (CRP) treatment components will be assessed and measured by ecological momentary assessments (EMA) between the treatment groups. EMA questions utilize a discrete rating scale to measure utilization of the treatment components.
Feasibility and acceptability of the experimental treatment as measured by qualitative interview. | Approximately 14 days post-intervention.
  The feasibility and acceptability of the experimental treatment will be measured by open-ended questions during a qualitative interview.
Changes in suicidal ideation, intent, behaviors, and urges as measured by ecological momentary assessments. | EMA surveys will be sent 5 times daily for 14 days pre-intervention and 5 times daily for 14 days post-intervention.
  Self-reported suicidal ideation, intent, behaviors, and urges will be repeatedly assessed throughout the protocol using ecological momentary assessments (EMA). EMA questions utilize a discrete rating scale to measure changes from pre-treatment and post-treatment.
Changes in thoughts of death and suicide as measured by the Ask Suicide-Screening Questions (ASQ) questionnaire. | Approximately 2 weeks before treatment and approximately 2 weeks after treatment.
  Self-reported thoughts of death and suicide will be assessed utilizing the Ask Suicide-Screening Questions (ASQ) questionnaire. The ASQ utilizes "yes" or "no" questions to assess thoughts of death and suicide "during the past few weeks".
Changes in suicidal ideation, intent, behaviors, and urges as measured by the Beck Scale for Suicidal Ideation (BSSI) questionnaire. | Approximately 2 weeks before treatment and approximately 2 weeks after treatment.
  Self-reported suicidal ideation, intent, behaviors, and urges will be assessed utilizing the Beck Scale for Suicidal Ideation (BSSI) questionnaire. Each question on the BSSI utilizes a rating scale of 0, 1, and 2 and a total score is calculated by summing the score for each question.
Changes in suicidal ideation, intensity, behaviors, and intent as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS). | Approximately 2 weeks before treatment and approximately 2 weeks after treatment.
  Suicidal ideation, intensity, behaviors, and intent will be assessed utilizing the Columbia-Suicide Severity Rating Scale (C-SSRS) interview. The C-SSRS interview utilizes "yes" or "no" questions. The C-SSRS also utilizes open-ended questions about how recently the thought or behavior occurred and the interviewer scores the severity based on a standard rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States